CLINICAL TRIAL: NCT03328858
Title: A Phase II Study of the Ketogenic Diet in Children With Malignant or Recurrent/Refractory Brain Tumor
Brief Title: Ketogenic Diet in Children With Malignant or Recurrent/Refractory Brain Tumor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer available, not able to find replacement. 2 patients, lost to follow-up.
Sponsor: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCH05817
Record Dates: First submitted 2017-10-23; First posted 2017-11-01 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Brain Tumors
Keywords: Ketogenic Diet, brain tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Ketogenic Diet will be initiated as inpatient, once all necessary studies are obtained and reviewed. The "classic ketogenic diet" will be initiated, and once ketosis is reached and patient demonstrates tolerance to diet he/she will be discharged home. Follow-up visits will be necessary up to 1 year.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic Diet (Other): Participants will be provided a consultation with a ketogenic dietitian, and test the tolerance to the diet in an inpatient mode
  Interventions: Other: Ketogenic Diet

INTERVENTIONS:
Other: Ketogenic Diet — Once tolerance to the diet has been assessed, participants will be placed in the ketogenic diet, followed-up every three months until the one year completion.

SUMMARY:
The purpose of this study is to evaluate the effect of the ketogenic diet on tumor size and quality of life in pediatric patients with malignant or recurrent/refractory brain tumors.

DETAILED DESCRIPTION:
Brain tumors account for nearly 20% of all childhood malignancies. Of these, gliomas represent 50% of all brain tumors in children and young adults. Gliomas are classically divided into two subtypes - low-grade and high-grade. Low-grade gliomas (LGG) include pilocytic astrocytomas and diffuse astrocytomas, and high-grade gliomas (HGG) include anaplastic astrocytoma and glioblastoma multiforme. Although patients with grade I and II tumors have a good prognosis with 5-year overall survival rates of 80-90%, those cases that are recurrent, refractory, and/or unresectable remain a challenge. The prognosis of children and young adults with recurrent or refractory malignant brain tumors remains poor despite dramatic improvements in treatment over the past few decades, with only a minority achieving long-term survival if recurrence occurs following initial surgical resection and adjuvant chemotherapy.

For patients with HGG prognosis remains dismal despite aggressive treatment. In this subset of patients, the 5-year overall survival for anaplastic astrocytoma ranges from 20-40% and for glioblastoma 15-20%. Diffuse intrinsic brain stem gliomas (DIPG) have the worst overall prognosis with a nine-month mean overall survival and with most patients dying from the disease within 2 years. Thus, the development of new treatment protocols for children and young adults with both high grade gliomas and with recurrent or refractory low grade gliomas is crucial to improving the survival rates of these patients.

The Ketogenic Diet (KD) has been in clinical use for nearly a century, initially designed to mimic the effects of starvation. Over the last two decades metabolic studies have been gaining momentum as increasingly promising in disease modification of central nervous system disorders and tumors.

Tests in animals and studies in adult patients with brain tumors have shown that there are advantages to using the ketogenic diet. These include: improved response of the tumor to standard treatment (chemotherapy/radiation) and improvement in quality of life measures (alertness).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis Medulloblastoma, high-grade glioma, low-grade glioma, and ependymoma are eligible. Other central nervous system tumors may be considered for treatment at discretion of investigator. Pathology is required unless diffuse intrinsic pontine glioma or optic pathway tumor. The patient should have failed first line therapy and be considered refractory, relapsed, or recurrent. Exceptions are Grade III and Grade IV gliomas including brain stem gliomas who can be enrolled at initial diagnosis.
* Prior Therapy Patients should have already had first line standard of care therapy, unless their initial diagnosis is high grade glioma or DIPG in which case they are eligible. Patients with high grade glioma can be enrolled after the completion of initial radiation. Investigator discretion may also be used.
* Organ Function Requirements A. Functioning gastrointestinal system, i.e. ability to chew and swallow or alternative means of nutrition therapy such as a gastrostomy or jejunostomy tube B. SGPT (ALT) < 3 x upper normal limit; Total Bilirubin ≤ 2 x upper normal limit C. No active pancreatitis D. No arrhythmia or prolonged QT.

Exclusion Criteria:

* History of cardiac arrhythmia
* Patient unable to chew/swallow and who do not consent to alternative methods of nutrition support, e.g. nasogastric or nasoduodenal tube, or gastrostomy or jejunostomy tube placement.

Ages: 12 Months to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | one year
  To evaluate the overall response rate of subjects with malignant or refractory brain tumors receiving dietary therapy with the ketogenic diet

SECONDARY OUTCOMES:
Quality of Life Measures | one year
  To evaluate the changes of quality of life of subjects with relapsed or refractory brain tumors receiving dietary therapy with the ketogenic diet using age-appropriate quality of life modules (Peds QL).
Ketosis Levels | one year
  To compare the betahydroxybutyrate level to decrease tumor size using MRI.
Blood Glucose Levels | one year
  To compare average blood glucose during ketogenic diet initiation compared to decrease in tumor size at time of first follow-up MRI.
Correlation of ketosis levels and ketogenic diet | one year
  To evaluate correlation between degree of ketosis (betahydroxybutyrate level) and ketogenic diet ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Caceres, MS, RDN, Principal Investigator — Nicklaus Children's Hospital; Ziad Khatib, MD, Study Director — Nicklaus Children's Hospital
Locations (1):
- Nicklaus Children's Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gasior M, Rogawski MA, Hartman AL. Neuroprotective and disease-modifying effects of the ketogenic diet. Behav Pharmacol. 2006 Sep;17(5-6):431-9. doi: 10.1097/00008877-200609000-00009. PMID 16940764
- [Background] Neal EG, Chaffe H, Schwartz RH, Lawson MS, Edwards N, Fitzsimmons G, Whitney A, Cross JH. A randomized trial of classical and medium-chain triglyceride ketogenic diets in the treatment of childhood epilepsy. Epilepsia. 2009 May;50(5):1109-17. doi: 10.1111/j.1528-1167.2008.01870.x. Epub 2008 Nov 19. PMID 19054400
- [Background] Kossoff EH. More fat and fewer seizures: dietary therapies for epilepsy. Lancet Neurol. 2004 Jul;3(7):415-20. doi: 10.1016/S1474-4422(04)00807-5. PMID 15207798
- [Background] Lussier DM, Woolf EC, Johnson JL, Brooks KS, Blattman JN, Scheck AC. Enhanced immunity in a mouse model of malignant glioma is mediated by a therapeutic ketogenic diet. BMC Cancer. 2016 May 13;16:310. doi: 10.1186/s12885-016-2337-7. PMID 27178315
- [Background] Vidone M, Clima R, Santorsola M, Calabrese C, Girolimetti G, Kurelac I, Amato LB, Iommarini L, Trevisan E, Leone M, Soffietti R, Morra I, Faccani G, Attimonelli M, Porcelli AM, Gasparre G. A comprehensive characterization of mitochondrial DNA mutations in glioblastoma multiforme. Int J Biochem Cell Biol. 2015 Jun;63:46-54. doi: 10.1016/j.biocel.2015.01.027. Epub 2015 Feb 7. PMID 25668474
- [Background] Nebeling LC, Miraldi F, Shurin SB, Lerner E. Effects of a ketogenic diet on tumor metabolism and nutritional status in pediatric oncology patients: two case reports. J Am Coll Nutr. 1995 Apr;14(2):202-8. doi: 10.1080/07315724.1995.10718495. PMID 7790697
- See also: Nicklaus Children's Hospital — https://www.nicklauschildrens.org/home